CLINICAL TRIAL: NCT05999786
Title: Effectivity of Early Recovery Accelerated Swallowing Program on Promoting Swallowing Recovery in Older Patients With High Risk of Oral Frailty Requiring Endotracheal Intubation During General Anesthesia: a Pilot Randomized Control Trial
Brief Title: ERAS Swallowing Rehabilitation in Elder Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Principal Investigator, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202303005RIND
Record Dates: First submitted 2023-08-06; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: The Upper Esophageal Sphincter Contraction Strength

STUDY DESIGN:
Intervention Model Description: Patients receive early recovery of swallowing rehabiliation before surgery and continued to after surgery
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data manager knows whether the patients are in the intervention or control group. However, the patients, caregiver, investigator, and outcome assessors do not know whether the patients are in the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients receiving early rehabiliation swallowing program (Active Comparator): the early rehabilitation program beginning from before to after surgery
  Interventions: Behavioral: early rehabiliation swallowing program
- patients not receiving early rehabilitation swallowing program (Placebo Comparator): the Taiwan Dysphagia Society's publicly shared swallowing exercises for dysphagia, which is started from before to after surgery
  Interventions: Behavioral: not receiving early rehabilitation swallowing program

INTERVENTIONS:
Behavioral: early rehabiliation swallowing program — not receiving early rehabilitation swallowing program from before and after surgery
  Arms: patients receiving early rehabiliation swallowing program
Behavioral: not receiving early rehabilitation swallowing program — the Taiwan Dysphagia Society's publicly shared swallowing exercises for dysphagia, which is from before and after surgery
  Arms: patients not receiving early rehabilitation swallowing program

SUMMARY:
The investigators studied that swallowing function of patients receiving the Early Recovery Accelerated Swallowing (ERAS-W program) training will recover fast than that of patients in the control group. The ERAS program training will be initiated before surgery and continue to after surgery.

DETAILED DESCRIPTION:
The older patients (≥65 years old) with OFI-8≥4 undergoing elective orthopedic surgery requiring tracheal intubation will be recruited. Patients will be randomized into an intervention and a control group. Patients in the intervention groups will received the ERAS-W program, while those in the control group will receive the swallowing education video.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery
* general anesthesia with endotracheal intubation

Exclusion Criteria:

* major organ dysfunction, ex: chronic kidney disease, hear failure
* bleeding tendency

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
UES pressure, mmHg | about six months

IPD SHARING:
Plan to Share IPD: No
due to ethical problem